CLINICAL TRIAL: NCT04756505
Title: REINA: A Phase I Study of Radiation Enhanced IL 12-Necrosis Attraction in Hormone Receptor Positive, HER2 Negative Metastatic Breast Cancer Patients
Brief Title: Immunotherapy (NHS-IL12 & Bintrafusp Alfa) and Radiation Therapy for the Treatment of Hormone Receptor Positive, HER2 Negative Metastatic Breast Cancer, the REINA Trial
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Per Sponsor Request-no longer manufacturing the study drug
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0245; NCI-2021-00434 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0245 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Hormone Receptor Positive Breast Adenocarcinoma; Metastatic Breast Carcinoma; Metastatic HER2 Negative Breast Adenocarcinoma; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms | interventions — bintrafusp alfa protein, human; NHS-IL12 immunocytokine; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (bintrafusp alfa, NHS-IL12, radiation therapy) (Experimental): Patients receive bintrafusp alfa IV over 1 hour on days 1 and 14 and immunocytokine NHS-IL12 SC on day 14. Beginning on day 14 of cycle 1, patients undergo radiation therapy QD for up to 4 days. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bintrafusp Alfa; Biological: Immunocytokine NHS-IL12; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Bintrafusp Alfa — Given IV
  Other Names: Anti-PDL1/TGFb Trap MSB0011359C; M7824; MSB0011359C
Biological: Immunocytokine NHS-IL12 — Given SC
  Other Names: M-9241; M9241; NHS-IL-12; NHS-IL12
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase I trial is to find out the best dose, possible benefits and/or side effects of NHS-IL12 given together with bintrafusp alfa and radiation therapy in treating patients with hormone receptor positive, HER2 negative breast cancer that has spread to other places in the body (metastatic). Immunotherapy with NHS-IL12, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Immunotherapy with bintrafusp alfa, a bifunctional fusion protein composed of the monoclonal antibody avelumab and TGF-beta, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving NHS-IL12, bintrafusp alfa, and radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of bintrafusp alfa (M7824) in combination with immunocytokine NHS-IL12 (NHS-IL-12) and radiation therapy in patients with metastatic hormone receptor positive (HR+)/HER2- breast cancer.

II. To determine the recommended phase II dose (RP2D) of NHS-IL-12 in combination with M7824 and radiation therapy in patients with metastatic HR+/HER2- breast cancer.

SECONDARY OBJECTIVES:

I. To assess immunologic/molecular responses, specifically percent (%) change in tumor infiltrating lymphocytes (TIL) pre and post therapy to M7824 in combination with NHS-IL-12 and radiation therapy in patients with HR+/HER2- metastatic breast cancer.

II. To explore preliminary progression free survival (PFS) and overall survival (OS) to power future definitive trial.

III. To evaluate the in-field and abscopal effect of treatment with M7824 in combination with NHS-IL-12 and radiation therapy.

EXPLORATORY OBJECTIVES:

I. To characterize circulating immune cell populations and cytokine profiles in tumor and circulation following treatment with M7824.

II. To conduct tissue-based ribonucleic acid sequencing (RNAseq), RNA scope, whole exome sequencing (WES) targeted sequencing.

III. To correlate dosimetry to response (assessed by degree of radiation fibrosis).

IV. To evaluate the pharmacokinetics of NHS-IL-12 in combination with M7824.

OUTLINE: This is a dose-escalation study of immunocytokine NHS-IL12.

Patients receive bintrafusp alfa intravenously (IV) over 1 hour on days 1 and 14 and immunocytokine NHS-IL12 subcutaneously (SC) on day 14. Beginning on day 14 of cycle 1, patients undergo radiation therapy once daily (QD) for up to 4 days. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Is willing and able to provide written informed consent for the trial and has signed the appropriate written informed consent form, approved by the investigator's Institutional Review Board (IRB)/Independent Ethics Committee (IEC), prior to the performance of any trial activities
* Is age >= 18 years at time of study entry
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Women of childbearing potential must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 8 weeks after the last dose of investigational product in such a manner that the risk of pregnancy is minimized. Men on study also must be using contraception. Women of childbearing potential (WOCBP) are women who have not been postmenopausal greater than 1 year or undergone a hysterectomy or bilateral oophorectomy
* Has confirmed HR+ and HER2 negative breast cancer with known metastatic disease. Eligible patients must have estrogen receptor (ER) and/or progesterone (PR) expression 10% or greater by immunohistochemistry (IHC). HER2 negative or nonamplified is determined by the current American Society of Clinical Oncology- College of American Pathologists (ASCO-CAP) criteria which are as follows: HER2 testing by IHC as 0 or 1+. If HER2 is 2+, ISH (in situ hybridization) must be performed. HER2 is positive if:

  * IHC 3+ based on circumferential membrane staining that is

    * Complete, intense
  * ISH positive based on:

    * Single-probe average HER2 copy number >= 6.0 signals/cell
    * Dual-probe HER2/CEP17 ratio >= 2.0 with an average HER2 copy number >= 4.0 signals/cell
    * Dual-probe HER2/CEP17 ratio >= 2.0 with an average HER2 copy number < 4.0 signals/cell
    * Dual-probe HER2/CEP17 ratio < 2.0 with an average HER2 copy number >= 6.0 signals/cell
* Has at least 2 identified sites of metastatic disease. This can include areas of metastatic disease to the bone, but one additional of the sites of metastatic disease must be amenable to biopsy
* Has measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Has received no more than 5 previous lines of chemotherapy and has received at least one line of therapy with an endocrine therapy or endocrine therapy combination
* Hemoglobin >= 10.0 g/dL
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (>= 1500 per mm^3)
* Platelet count >= 100 x 10^9/L (>= 100,000 per mm^3)
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only upon treating physician, principle investigator (PI) or co-PI approval
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be =< 5 x ULN
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits, examinations, and assessments (including follow up)
* Protocol participation is such that the treatment will be administered as an outpatient. Inpatient status is not required and change in status does not necessitate removal from protocol
* Has not had major surgery within 28 days prior to starting study treatment. Central venous access surgeries and/or placements would not be considered as major surgery

Exclusion Criteria:

* Anticancer treatment within 14 days before the start of trial treatment (e.g. cytoreductive therapy, radiotherapy etc.), or surgery within 4 weeks of start of trial treatment
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease =< 3 years before the first dose of study drug and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease eg, cervical cancer in situ
* QT interval corrected for heart rate (QTc) >= 470 ms
* Current or prior use of immunosuppressive medication within 28 days before the first dose of M7824 or NHS-IL-12, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
* Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, hypo- or hyperthyroid disease, or psoriasis not requiring systemic treatment are not excluded
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* Significant acute or chronic infections including, among other:

  * Known history of testing positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome
  * Active hepatitis B virus (HBV surface antigen positive) or hepatitis C virus (HCV antibody positive and/or HCV RNA positive)
  * Subjects with known active tuberculosis (history of exposure or history of positive tuberculosis test plus presence of clinical symptoms, physical or radiographic findings)
* History of allogeneic organ transplant
* History of hypersensitivity to M7824 or NHS-IL-12 or any excipient of either compound
* History of uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of a psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* Known history of previous clinical diagnosis of tuberculosis
* Subjects with active central nervous system (CNS) metastases causing clinical symptoms or metastases that require therapeutic intervention, including leptomeningeal disease, are excluded. Subjects with a history of treated CNS metastases (by surgery or radiation therapy) are not eligible unless they have demonstrated no progression for at least 1 month, and do not require continued steroid therapy.
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving study drugs
* Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control
* Any condition, including chronic medical condition, that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
* Subjects with uncontrolled seizures
* Any absolute contraindication to protocol specified radiotherapy based on prior radiotherapy (determined by radiation oncologist)
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti- Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways) for metastatic breast cancer. Or, if patient has had prior immune-oncology therapies in the neoadjuvant or adjuvant setting within the past 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-07 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days post treatment
  Detailed information collected for each AE will include a description of the event, duration, severity, relationship to study treatment, action taken and clinical outcome. Severity of AEs will be grated according to Common Terminology Criteria for Adverse Events version .4.0.
Recommended phase II dose (RP2D) | Up to 28 days
  RP2D will be determined by "3+3" design, and the recommended phase II dose is defined when 6 patients have been treated on that dose with no more than 1 dose-limiting toxicity.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From start of treatment until objective tumor progression or death, whichever occurs first, assessed up to 1 year
  PFS will be estimated for all enrolled patients and patients who receive at least one treatment using Kaplan-Meier method and compared between or among patients' characteristic groups by log-rank test. Univariate Cox regression model may be applied to assess the effect of variables of interest on PFS when appropriate.
Overall survival (OS) | From treatment until death from any cause, assessed up to 1 year
  OS will be estimated for all enrolled patients and patients who receive at least one treatment using Kaplan-Meier method and compared between or among patients' characteristic groups by log-rank test. Univariate Cox regression model may be applied to assess the effect of variables of interest on OS, when appropriate.
Percent (%) change in tumor infiltrating lymphocytes (TIL) | Baseline up to 1 year
  The % change of TIL pre and post treatment will be estimated along with 95% confidence interval. Wilcoxon signed rank test may be used to examine whether the change in TIL is different from zero.
Size of metastasis after treatment with both therapeutic agents with radiation (in-field) and nonirradiated (abscopal) sites | Up to 1 years
  The difference in size of metastasis measured by the longest diameters of the tumor or the shortest diameter of a lymph node by Response Evaluation Criteria in Solid Tumors, before and after treatment will be estimated for both the irradiated site (diff irradiated) and the non-irradiated site (diff non-irradiated). Will also estimate the difference between the two different sites (diff = diff non-irradiated - diff irradiated). May evaluate if diff irradiated, diff non-irradiated, and diff = diff non-irradiated - diff Irradiated are significantly different from 0 by the Wilcoxon signed rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Karuturi, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org